CLINICAL TRIAL: NCT01791426
Title: A Study to Evaluate the Performance and Safety of Artelac Rebalance® Versus Vismed in the Management of Dry Eye
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Adjustment of company focus due to acquision by Valeant Pharmaceuticals
Sponsor: Bausch & Lomb Incorporated (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single
Other Study IDs: 810
Record Dates: First submitted 2013-02-04; First posted 2013-02-15 (Estimated); Last update posted 2013-10-11 (Estimated); Status verified 2013-10

CONDITIONS: Dry Eye
MeSH Terms: conditions — Dry Eye Syndromes

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Artelac Rebalance (Experimental): Artelac Rebalance ophthalmic solution contains 0.15% hyaluronic acid, is unpreserved and presented in single dose units with a fill volume of 0.5 mL.
  Interventions: Device: Artelac Rebalance
- Vismed (Active Comparator): Vismed ophthalmic solution, contains 0.18% sodium hyaluronate, is unpreserved and presented in single dose units with a fill volume of 0.3 mL.
  Interventions: Device: Vismed

INTERVENTIONS:
Device: Artelac Rebalance — Instill 1 drop of the Artelac Rebalance eye drops in each eye 3 to 5 times per day for 90(± 10) day treatment.
  Arms: Artelac Rebalance
Device: Vismed — Instill 1 drop of the Vismed eye drops in each eye 3 to 5 times per day for 90(± 10) day treatment.
  Arms: Vismed

SUMMARY:
The objective of this investigation is to show that the performance of Artelac Rebalance eye drops is non-inferior to that of Vismed eye drops in subjects with moderate to severe dry eye, and to assess the safety of Artelac Rebalance after a 90-day (± 10 day) treatment administered 3 to 5 times per day.

DETAILED DESCRIPTION:
Artelac Rebalance and Vismed are in compliance with European Directives (CE marked) products in the European Union (EU).

ELIGIBILITY:
Inclusion Criteria:

* Subjects who have been using tear substitutes for at least 3 months prior to inclusion, and who will use preservative-free ART (Artelac® UNO CL hypromellose 0.32% w/v eye drops, single dose unit) up to 6 times a day for at least 2 weeks immediately prior to randomization
* Subjects with at least 1 eye with the following signs of keratoconjunctivitis sicca at 2 consecutive visits (Visit 1[Screening] and Visit 2 [Randomization])
* Schirmer test without anesthesia of ≤ 9 mm/5min
* Tear break-up time of ≤ 10sec (mean of 3 measurements)
* Total ocular surface staining score ≥ 4 and ≤ 9. This assessment combines corneal fluorescein staining and nasal and temporal bulbar conjunctival lissamine green staining, each graded 0-5 according to the Oxford Scheme
* Subjects who have a decimal visual acuity (VA) with habitual correction equal to or better than 0.1 (Snellen E chart) in both eyes
* Subjects who are receiving stable systemic treatment (unchanged for 1 month or longer)

Exclusion Criteria:

* Subjects with moderate or severe blepharitis
* Subjects who have severe ocular dryness accompanied by 1 of the following:
* Lid abnormality (except mild blepharitis)
* Corneal disease
* Ocular surface metaplasia
* Filamentary keratitis
* Corneal neovascularization
* Subjects who currently wear contact lenses or have worn contact lenses within 90 days prior to study start
* Subjects who have received ocular surgery, including laser surgery, in either eye within 180 days prior to study start
* Subjects with a history of ocular trauma, non-dry eye ocular inflammation, or ocular infection within 90 days prior to study start
* Subjects with a history of ocular allergic disease or ocular herpes within

  1 year prior to study start
* Subjects with a history of any inflammatory ulcerative keratitis, recurrent corneal erosion, or uveitis
* Subjects with known hypersensitivity or contraindications to any of the ingredients in the test or comparator products
* Subjects with planned initiation of, or changes to, concomitant medication that could affect dry eye within 30 days of Visit 1 (Screening) or during the study
* Subjects who have received ocular therapy (either eye) with any ophthalmic medication, except tear substitutes, within 2 weeks prior to study start
* Subjects expected to receive ocular therapy during the study
* Subjects treated with topical ocular steroidal or non-steroidal anti- inflammatory medication within 30 days prior to study start
* Subjects expected to receive ocular therapy with immunosuppressants (eg, cyclosporine) during the study or who have used ocular immunosuppressants within 90 days prior to study start
* Subjects who have received occlusion therapy with lacrimal or punctum plugs within 90 days prior to study start

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2013-05; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

PRIMARY OUTCOMES:
Combined Ocular Surface Staining Score | Mean change from baseline (CFB) to visit 4 (day 28)
  Total combined ocular surface staining grade of 0-15 combining corneal fluorescein staining score, nasal and temporal bulbar conjunctiva lissamine green staining score (each graded 0-5 on the Oxford Scheme) in the study eye.

SECONDARY OUTCOMES:
Combined Ocular Surface Staining Score | Mean CFB to visit 3 (Day 7) visit 4 (Day 28) and visit 5 (Day 90)
  Mean CFB in the study eye at Visits 3, 4 and 5 in total combined ocular surface staining score.
Corneal Fluorescein Staining Score | Mean CFB at each follow-up visit: visit 3 (Day 7) visit 4 (Day 28) and visit 5 (Day 90)
  Mean CFB in the study eye in corneal fluorescein staining score at each follow-up visit
Nasal Conjunctival Lissamine Green Staining | Mean CFB at each follow-up visit: visit 3 (Day 7) visit 4 (Day 28) and visit 5 (Day 90)
  Mean CFB in the study eye in nasal conjunctival lissamine green staining at each follow-up visit.
Temporal Conjunctival Lissamine Green Staining | Mean CFB at each follow-up visit: visit 3 (Day 7) visit 4 (Day 28) and visit 5 (Day 90)
  Mean CFB in the study eye in temporal conjunctival lissamine green staining at each follow-up visit
Tear Film Break-up Time | Mean CFB at each follow-up visit: visit 3 (Day 7) visit 4 (Day 28) and visit 5 (Day 90)
  Mean CFB in the study eye in tear film break-up time (TFBUT) at each follow-up visit.
Study Drop Sensation | Each follow-up visit: visit 3 (Day 7) visit 4 (Day 28) and visit 5 (Day 90)
  Study drop sensation, as reported by subject in subject diary

CONTACTS AND LOCATIONS:
Overall Officials: Helmut Allmeier, PhD, Study Director — Bausch & Lomb Incorporated